CLINICAL TRIAL: NCT01987557
Title: The Therapeutic Contributions of Somatosensory Feedback During Exercise in Parkinson's Disease; A Randomized, Controlled Trial.
Brief Title: Amplitude and Rate of Intrinsic Feedback During Treadmill Training for Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wilfrid Laurier University (Other)
Responsible Party: Principal Investigator, Matthew Lasswell, Mr. Matthew Lasswell, Wilfrid Laurier University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MDRC
Record Dates: First submitted 2013-10-09; First posted 2013-11-19 (Estimated); Results first posted 2015-06-17 (Estimated); Last update posted 2015-06-17 (Estimated); Status verified 2015-06

CONDITIONS: Parkinson's Disease; Treadmill
Keywords: treadmill; parkinson's; proprioception; cadence; step length; intrinsic feedback
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Treadmill Intervention 1: Rate Group (Experimental): Participants in this condition will walk with a cadence (steps per minute) that is approximately 35% faster than comfortable walking pace. In this condition, participants will maintain a step length that is similar to that of their comfortable walking pace.
  Interventions: Behavioral: rate group
- Magnitude treadmill group (Experimental): In this condition participants will walk on a treadmill with weights on their ankles to elicit a greater magnitude of instrinsic feedback from force sensitive golgi tendon organs
  Interventions: Behavioral: magnitude treadmill group
- regular treadmill walking (Placebo Comparator): participants will walk at a comfortable self-selected pace on a treadmill
  Interventions: Behavioral: regular treadmill walking

INTERVENTIONS:
Behavioral: rate group — walking with a high cadence (steps per minute)
  Arms: Treadmill Intervention 1: Rate Group
Behavioral: magnitude treadmill group
  Arms: Magnitude treadmill group
Behavioral: regular treadmill walking
  Arms: regular treadmill walking

SUMMARY:
Treadmill training has been shown to be beneficial for reducing motor symptoms of Parkinson's disease (PD). The mechanisms for the therapeutic effects of treadmill training remain unknown. However, specific types of intrinsic feedback generated from muscle spindles (detect changes in length of muscle) and golgi tendon organs (detect muscle force) seem to be an important factor for achieving the reductions in motor scores. This study will compare a treadmill program that generates a high rate of intrinsic feedback to a treadmill program focused on generating a high magnitude of intrinsic feedback.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of Parkinson's disease
* must be able to walk unassisted for 10 metres

Exclusion Criteria:

* cardiovascular disease/history of stroke
* Dementia
* lower body injury that would be worsened by repetitive walking

Ages: 40 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2013-10; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

RESULTS

PARTICIPANT FLOW:
Groups:
- Magnitude Treadmill Group: In this condition participants will walk on a treadmill with weights on their ankles to elicit a greater magnitude of instrinsic feedback from force sensitive golgi tendon organs
  magnitude treadmill group
- Regular Treadmill Walking: participants will walk at a comfortable self-selected pace on a treadmill
  regular treadmill walking
Period: Overall Study
Arm/Group | Treadmill Intervention 1: Rate Group | Magnitude Treadmill Group | Regular Treadmill Walking
Started | 16 | 16 | 16
Completed | 13 | 13 | 13
Not Completed | 3 | 3 | 3
Not completed — Protocol Violation | 1 | 0 | 1
Not completed — Withdrawal by Subject | 2 | 1 | 2
Not completed — Adverse Event | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treadmill Intervention 1: Rate Group | Magnitude Treadmill Group | Regular Treadmill Walking | Total
Number analyzed (Participants) | 13 | 13 | 13 | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.77 (7.01) | 70.46 (9.52) | 66.31 (9.07) | 66.85 (8.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 1 | 5
  Male | 10 | 12 | 12 | 34
Unified Parkinsons Disease Rating Scale-Motor Subsection (UPDRS III) [Mean (Standard Deviation); unit: units on a scale] | 23.35 (8.13) | 22.96 (6.93) | 22.46 (8.64) | 22.92 (7.73)

OUTCOME MEASURES:

1. Primary Outcome: Motor Section of the Unified Parkinson's Disease Rating Scale (UPDRS-III)
Description: A measure of the motor symptom severity within Parkinsons. UPDRS III is a qualitative assessment performed by a trained clinician. Specifically, a change in UPDRS III from pre to post is the main outcome measure.
  The UPDRS-III score is a summation of 27 tasks that are scored from 0-4. 0 meaning no impairment, and 4 representing extreme impairment, inability to complete task. Possible scores on the UPDRS-III range from 0 (no impairment) to 108 (extreme impairment).
Time Frame: Pre assessments are conducted in the week prior to the treadmill program. Post are conducted during the week immediately following the program. Changes after the 6 week treadmill program are being examined
Measure: Mean (Standard Deviation); unit: units on a scale (0-4)
Arm/Group | Treadmill Intervention 1: Rate Group | Magnitude Treadmill Group | Regular Treadmill Walking
Number analyzed (Participants) | 13 | 13 | 13
units on a scale (0-4)
  PRE | 23.35 (8.13) | 22.96 (6.93) | 22.46 (8.64)
  POST | 18.81 (7.17) | 20.69 (8.39) | 20.92 (6.14)

2. Secondary Outcome: Spatiotemporal Aspects of Gait
Description: Participants will walk on a pressure sensitive GAITRite carpet (Sparta, NJ), at both comfortable and fast paced walking speeds. Changes in gait characteristics from pre to post are what is being examined.
  Quantitative measures of gait such as step time, step length, walking velocity, and others will be used in the analysis.
  Spotters are always present to ensure safety during this assessment.
Time Frame: pre test occurs within the week prior to the start of the treadmill training program. Post testing will occur during the week immediately following the 6 week treadmill training program.
Reporting Status: Not Posted

3. Secondary Outcome: Static Posturography (Balance/Postural Control)
Description: A Balance SD system from BIODEX (Shirley, NY) will be used to assess postural control. Changes from pre to post are what is being examined.
Time Frame: as for outcome 2
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Treadmill Intervention 1: Rate Group | Magnitude Treadmill Group | Regular Treadmill Walking
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 0/16 | 2/16 | 0/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treadmill Intervention 1: Rate Group (N=16) | Magnitude Treadmill Group (N=16) | Regular Treadmill Walking (N=16)
Muscle Strain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) — Mild Hamstring strain.
back muscle tightness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) — minor back muscle discomfort leading the participant withdraw from the study

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes